CLINICAL TRIAL: NCT04990323
Title: A Phase I/II Open-Label Study of ECT-001-Expanded Cord Blood Transplantation in Pediatric and Young Adult (<21year) Patients With High-Risk and Very High-Risk Myeloid Malignancies
Brief Title: US Study of ECT-001-CB in Pediatric and Young Adult Patients With High-Risk Myeloid Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ExCellThera inc. (Industry)
Collaborators: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECT-001-CB.007
Record Dates: First submitted 2021-07-27; First posted 2021-08-04 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: High Risk Myeloid Malignancies; Cord Blood Transplant
MeSH Terms: interventions — Transplantation Conditioning; Cyclophosphamide; Thiotepa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ECT-001-Expanded CB (Experimental): Patients will receive a myeloablative conditioning regimen (Preferred: Clo/Flu/Bu90, Alternative: MIDI)
  The cord to be expanded will undergo CD34+ selection. The CD34- product is cryopreserved and will be thawed and infused on Day +1 post-transplant. The CD34+ product will be placed in a closed culture with UM171 for a 7-day expansion and is infused on Day 0.
  Patients will receive standard supportive care and GVHD prophylaxis (such as MMF and tacrolimus).
  Interventions: Biological: ECT-001-CB (UM171-Expanded Cord Blood Transplant)

INTERVENTIONS:
Biological: ECT-001-CB (UM171-Expanded Cord Blood Transplant) — Single UM171-Expanded CB transplant (CD34+: 2.5-50x10^5/kg, CD3+>1x10^6/kg)
  Other Names: Conditioning Regimen (Preferred): clofarabine:30 mg/m2/day IV x 4 days, fludarabine:10 mg/m2/day IV x 4 days, busulfan: daily for 4 days with cumm Bu target = 90mg h/L; Conditioning Regimen (Alternative): MIDI: fludarabine: 30 mg/m2/day IV x 5 days, cyclophosphamide: 50 mg/kg IV , thiotepa: 5 mg/kg/day IV x 2 days , TBI: 400 cGy; GVHD Prophylaxis: Tacrolimus/MMF

SUMMARY:
Cord blood (CB) transplants are an option for patients lacking an HLA identical donor but are hampered by low cell dose, prolonged aplasia and high transplant related mortality. UM171, a novel and potent agonist of hematopoietic stem cell self renewal could solve this major limitation, allowing for CB's important qualities as lower risk of chronic GVHD and relapse to prevail. In previous trials (NCT02668315, NCT03913026, NCT04103879, and NCT03441958), the CB expansion protocol using the ECT-001-CB technology (UM171 molecule) has proven to be technically feasible and safe in adults.

UM171 expanded CB was associated with a prompt (D+17), robust (98%) and durable neutrophil recovery. Amongst patients who received a single UM171 CB transplant with a median follow-up of 18 months, risk of TRM (10%), grade 3-4 acute GVHD (13%) and moderate-severe chronic GVHD (2%) was low at 1 year post-transplant. Incidence of severe viral and bacterial infections was reduced and immunosuppression could be discontinued in 77% of patients at 1 year. Thus, PFS and GRFS were very promising, 72% and 59% at 12 months, 69% and 53% at 24 months, respectively, in particular accounting for a large proportion of very high-risk patients. By a 10-fold increase of CB accessibility, ECT-001-CB allowed access to smaller, better HLA matched CBs.

This new study seeks to test a similar strategy in a group of pediatric and young adult patients with high risk myeloid malignancies. 12 patients will be enrolled in the first stage of this 2-stage design protocol. If intervention is considered promising (<= 3 relapses in the first 12 patients), this study will open multicenter and be extended to a second stage (16 additional patients for a total accrual 28).

ELIGIBILITY:
Inclusion Criteria:

1. Acute Myeloid Leukemia

   1. Chemo-refractory relapse (MRD+)
   2. Primary induction failure (no CR or CRi after >= 2 courses of intensive induction therapy): < 30% blasts in evaluable marrow.
   3. Relapse after previous allogeneic (or autologous) transplant (>4 months)
   4. Secondary or therapy-related MDS/AML
   5. Poor response to induction (5-30% blasts) or MDR+ after induction
2. Myelodysplastic syndrome (MDS)

   1. Relapse after allogeneic or autologous transplant (>4 months)
   2. ≥10 % blasts within 30 days of start of conditioning regimen
   3. Poor and very poor cytogenetics abnormalities
3. Chronic myelogenous leukemia: Patients who progressed to blast crisis
4. Mixed Phenotype Acute Leukemia: MRD+ or relapse after previous transplant (>4 months).
5. JMML (Juvenile Myelo-Monocytic Leukemia)
6. Availability of 2 ≥ 4/8 HLA matched CBU (allele level: A, B, C and DRB1)

   1. Cord to be expanded: CD34+ cell count ≥ 0.5 x 10^5/kg and TNC ≥ 1.5 x 10^7/kg (pre-cryo)
   2. Back up cord: Pre-freeze TNC ≥ 2 x 10^7/kg with CD34+ cells ≥ 1.5 x 10^5/kg. If a single cord does not meet this criterion 2 back up cords will be an acceptable alternative with a minimum for each of 1.5 x 10^7 TNC/kg with 1.0 x 10^5 CD34+/kg. Another acceptable HSC back up source could be a haploidentical with medical clearance prior to starting conditioning regimen.
7. Lansky / Karnofsky >60%
8. Bilirubin < 2 x upper limit of normal (ULN) unless felt to be related to Gilbert's disease or hemolysis; AST and ALT < 3 x ULN; alkaline phosphatase < 5 x ULN
9. Estimated or measured creatinine clearance ≥ 50ml/min/1.73m2
10. Left ventricular ejection fraction of ≥ 40%
11. FVC, FEV1 and DLCO ≥ 50% of predicted
12. Signed written informed consent
13. Female patients of childbearing potential must have a negative serum pregnancy test within 7 days of enrolment and mush be willing to use an effective contraceptive method while enrolled in the study.

Exclusion Criteria:

1. Previous allogeneic transplantation within 4 months.
2. Uncontrolled infection.
3. Presence of other malignancy other than the one for which the CB transplant is being performed, with an expected survival to be less than 75% at 5 years
4. Seropositive for HIV.
5. Hep B and C infection with measurable viral load.
6. Liver cirrhosis.
7. Active CNS disease.
8. Chloroma > 2cm.
9. >30% blasts in marrow in evaluable marrow sample.
10. Pregnancy, breastfeeding, or unwillingness to use appropriate contraception
11. Participation in a trial with an investigational agent within 30days prior to entry in the study.
12. Any abnormal condition or lab result that is considered by the PI capable or altering patient's condition or study outcome.

Ages: 0 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events of ECT-001-CB | 100 days
  Incidence and severity of AEs according to the modified (for HSCT) CTCAE (v. 5.0)
Relapse | 1 year post-transplant
  Incidence of relapse will be measured from time of transplant

SECONDARY OUTCOMES:
Leukemia-free survival | 1- and 2-year post-transplant
  LFS will be measured from time of transplant until disease relapse, death or last follow-up
Non-Relapse Mortality | 1 year post-transplant
  NRM is defined as any death of any cause other than malignant relapse, occurring after the commencement of conditioning regimen that could be related to the transplantation procedure
GVHD | 1- and 2-year post-transplant
  Incidence of acute and chronic GVHD will be measured by NIH criteria
Grade 3 Infections | 2-year post-transplant
  Incidence and severity of infections requiring systemic therapy, e.g., invasive candidiasis, aspergillus, other invasive fungi, CMV, adenovirus, EBV, HHV-6, HSV, VZV, PCP, toxoplasmosis and mycobacterium
Hematologic engraftment | 42 and 100 days
  Time to neutrophil engraftment (the first day of attainment of an absolute neutrophil count ≥0.5 x 10E9/L for 3 consecutive days. Time to ANC ≥ 0.1 x 10E9/L will also be documented) and time to platelet engraftment (first day of a sustained platelet count ≥ 50 x 10E9/L with no platelet transfusion in the preceding 7 days)
Pre-engraftment/engraftment syndrome | 2-year post-transplant
  Incidence of pre-engraftment/engraftment syndrome requiring therapy
Hospitalization events | 100 days
  Duration of transplant admission and number of days in hospital in 1st 100 days, and last day of fever (>38°C) prior to engraftment

CONTACTS AND LOCATIONS:
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR